CLINICAL TRIAL: NCT01177527
Title: Medical Questionnaire and Tissue Banking For Multiple Myeloma, Waldenstrom Macroglobulinemia and Related Disorders
Brief Title: Questionnaire and Tissue Banking For Multiple Myeloma, Waldenstrom Macroglobulinemia and Related Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 09-233
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Waldenstrom's Macroglobulinemia; Smoldering Multiple Myeloma; Lymphoblastic Lymphoma
Keywords: Waldenstrom; myeloma; smoldering; lymphoma; MGUS; distinct B-cell lymphoproliferative disorder
MeSH Terms: conditions — Multiple Myeloma; Waldenstrom Macroglobulinemia; Smoldering Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms, Plasma Cell; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood Bone marrow samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to obtain bone marrow and peripheral blood samples, along with clinical data from patients with Multiple Myeloma (MM), Waldenstrom's Macroglobulinemia (WM), Smoldering MM, and other lymphoplasmacytic lymphomas (LPL) including but not limited to MGUS and IgG or IgA LPL. These samples will become part of a tissue bank and will be used in ongoing studies to find out more about the causes and biology of MM, WM and LPL; to identify what factors result in normal cells becoming cancer; to determine how to improve treatment options; to study how the immune system identifies abnormal cells; and to evaluate the immune function in these diseases. The investigators will also study the tumor cells at the level of the participant's genes to develop treatment strategies as well as to better understand how biologic differences affect patient outcomes.

DETAILED DESCRIPTION:
* Participants will be asked to complete a medical survey which includes demographics, diagnosis, and treatment history, medical history, lab results and symptoms experienced.
* Participants will then receive instructions for the tissue banking procedure, which involves donating bone marrow and blood samples. These will be collected only at times when necessary clinical bone marrow samples are obtained and will not require an extra visit to the doctor.
* The investigators are also requesting permission to collect medical information from the participant's record and link this information to the specimens so that we may better understand the participant's response to treatment. For samples obtained prior to beginning therapy, this information might allow us to develop new ways of predicting response to therapy. The investigators are also requesting permission to store samples of blood and bone marrow to establish a tissue bank for future research to these diseases. These samples will be de-identified; any of the participant's personal health information identifiers will be removed.
* The tumor sample may be obtained at diagnosis, during treatment and/or as the time of relapse. The timing of sample collection will coincide with other bone marrow tests required to assess the response to therapy or any other clinical purpose.

ELIGIBILITY:
Inclusion Criteria:

* Any individual diagnosed with Multiple Myeloma, Waldenstrom Macroglobulinemia, MGUS, smoldering MM or other lymphoplasmacytic lymphomas
* Signed informed consent
* 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant's will be identified through several mechanisms:
  1. Primary recruitment will occur via Internet advertising through patient websites including but not limited to the International Waldenstrom's Macroglobulinemia Foundation (IWMF), the Leukemia and Lymphoma Society and the Multiple Myeloma Research Foundation (MMRF) websites.
  2. Investigators who identify patients at Dana-Farber Cancer Institute (DFCI) who do not wish to continue their treatment plan at DFCI can approach these patients to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 656 (Actual)
Dates: Start 2009-12; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Databank | 3 years
  To establish a databank of patients with MM, WM, MGUS, sMM, or related disorders. This databank will include medical history data and bone marrow and peripheral blood samples.
Unique characteristics | 3 years
  To determine whether patients with MM, WM, MGUS, sMM, or related disorders have unique proteomic, genetic and epigenetic characteristics in the malignant clone or the microenvironment and linking information to the clinical characteristics of the patients through exploratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States